CLINICAL TRIAL: NCT00693524
Title: An Open, Randomized, Multicentre Clinical Study to Compare the Safety and Efficacy of a Combination of Sequential Therapy of Tacrolimus (FK506) With Monoclonal Anti-IL2R Antibodies and Mycophenolate Mofetil Versus Tacrolimus (FK506) With Steroids in Liver Allograft Transplantation
Brief Title: Sequential Therapy (FK506 + Monoclonal Anti-IL2R Antibodies + MMF) Versus FK506 With Steroids in Liver TX
Acronym: TAST
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FG-506-01-IT-01
Record Dates: First submitted 2008-06-04; First posted 2008-06-09 (Estimated); Last update posted 2014-08-26 (Estimated); Status verified 2014-08

CONDITIONS: Liver Transplantation
Keywords: liver allograft transplantation; sequential therapy; tacrolimus
MeSH Terms: interventions — Tacrolimus; Daclizumab; Mycophenolic Acid; Prednisone; Steroids

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Tacrolimus + Anti-IL2R AB + Mycophenolate mofetil
  Interventions: Drug: tacrolimus; Drug: Anti-IL2R AB; Drug: Mycophenolate mofetil
- 2 (Active Comparator): Tacrolimus + Steroid
  Interventions: Drug: tacrolimus; Drug: prednisone

INTERVENTIONS:
Drug: tacrolimus — oral
  Other Names: FK506; Prograf
Drug: Anti-IL2R AB — i.v.
  Other Names: daclizumab
  Arms: 1
Drug: Mycophenolate mofetil — oral
  Arms: 1
Drug: prednisone — oral
  Other Names: steroid
  Arms: 2

SUMMARY:
Study to evaluate the benefits and any risks of the delayed administration of tacrolimus in a combined regimen of mycophenolate mofetil and monoclonal anti-IL2R antibodies (daclizumab), in comparison with a standard steroid + tacrolimus double drug regimen

ELIGIBILITY:
Inclusion Criteria:

* Patient is undergoing orthotopic liver allograft transplantation. This includes partial organ transplantation. Age of donor between 5 and 65 years

Exclusion Criteria:

* Patient has previously received or is receiving an organ transplant (including liver re-transplantation)
* Recipient of an auxiliary graft or in which a bio-artificial liver has been used
* Patient is receiving a living related liver transplantation
* Patient is requiring steroids as well as chemotherapy prior to transplantation
* Patient having any previous history of neoplastic disease of any type (including leukaemia). However, patients with primary liver carcinoma can be included if they meet the following criteria:

  * > 3 nodes
  * No node larger than 5 cm
  * No metastases
  * No vascular invasion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2002-11; Primary Completion 2004-03 (Actual); Study Completion 2004-03 (Actual)

PRIMARY OUTCOMES:
Incidence of first acute rejection | 3 months

SECONDARY OUTCOMES:
Overall frequences of acute rejection episodes | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Central Contact, Study Director — Astellas Pharma Europe B.V.
Locations (8):
- Italy (8):
  - Bologna
  - Genova
  - Milan
  - Napoli
  - Padua
  - Roma
  - Torino
  - Udine